CLINICAL TRIAL: NCT06848959
Title: Jiangsu Provincial Hospital of Traditional Chinese Medicine
Brief Title: Development and Application of a Diagnosis and Treatment System for Children's Brain Diseases Based on Knowledge Graphs and Large Models
Status: Recruiting | Type: Observational
Sponsor: Yun Liu,PhD (Other)
Responsible Party: Sponsor-Investigator, Yun Liu,PhD, PhD, Affiliated Hospital of Nanjing University of Chinese Medicine
Organization: Affiliated Hospital of Nanjing University of Chinese Medicine (Other)
Other Study IDs: HospitalNanjingU; Nanjing Science and Technology (Other: HospitalNanjingU)
Record Dates: First submitted 2025-02-18; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Palsy; Mental Retardation; Tourette's Syndrome; Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorders
MeSH Terms: conditions — Cerebral Palsy; Intellectual Disability; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — Pediatric Encephalopathy Science and Prevention Decision Aid Follow-Up Q&A

SUMMARY:
Using the knowledge graph and big model technology of combining Chinese and Western medicine we construct a popularization and prevention system for childhood encephalopathy an assisted decision-making system for childhood encephalopathy and a follow-up tracking question and answer system for childhood encephalopathy patients.

ELIGIBILITY:
Inclusion Criteria:

* 1. meet diagnostic criteria for CP ID TD ADHD ASD; 2. gender is not limited;

Exclusion Criteria:

* 1. CP ID TD ASD due to chorea hepatomegaly hearing abnormality and pharmacogenetic factors;
* 2. Children with other major mental illnesses (e.g. schizophrenia) or organic diseases (e.g. congenital heart disease);

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Childhood encephalopathy
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Childhood Autism Rating Scale | 4 mouths
  The total score ranges from 15 to 60, with the higher the score the worse the symptoms are
meridian and acupointological features | 4 mouths
  After obtaining the information through diagnosis by a professional Chinese medicine practitioner, assist in the diagnosis of clinical subtypes of children according to the corresponding typology of "Pediatrics of Chinese Medicine".
Yale Global Tic Severity Scale | 4 mouths
  It has a score range of 0-100, with higher scores representing more severe symptoms.
Gross Motor Function Assessment Scale (GMFM)-88 | 4 mouths
  GMFM-88 scores range from 0-264, with higher scores being better.
Autism Behavior Checklist | 4 mouths
  It has a score range of 0-174, with higher scores representing more severe symptoms.
acupuncture point status | 4 mouths
  After obtaining the information through diagnosis by a professional Chinese medicine practitioner, assist in the diagnosis of clinical subtypes of children according to the corresponding typology of "Pediatrics of Chinese Medicine".
Tongue texture | 4 mouths
  After obtaining the information through diagnosis by a professional Chinese medicine practitioner, assist in the diagnosis of clinical subtypes of children according to the corresponding typology of "Pediatrics of Chinese Medicine".
Wechsler intelligence scale (WIS) | 4 mouths
  FIQ = 100: Indicates that the individual has an average level of intelligence. FIQ > 100: Indicates an above average level of intelligence. FIQ < 100: Indicates a below average level of intelligence.
Resting heart rate | 4 mouths
blood pressure (systolic, diastolic) after 10 minutes of rest | 4 mouths
Conners Rating Scales | 4 mouths
  Scores are converted to standardized T-scores for comparison with the mean of the peer group. T-scores above 65 are usually considered clinically significant.
tongue coating, pulse | 4 mouths
  After obtaining the information through diagnosis by a professional Chinese medicine practitioner, assist in the diagnosis of clinical subtypes of children according to the corresponding typology of "Pediatrics of Chinese Medicine".
respiratory rate | 4 mouths
Body temperature | 4 mouths

SECONDARY OUTCOMES:
Saliva | 4 mouths
  Destruction after use. Metabolomics after sample collection.
blood | 4 mouths
  Destruction after use. Metabolomics after sample collection.
Urine | 4 mouths
  Destruction after use. Metabolomics after sample collection.
Faeces | 4 mouths
  Destruction after use. Metabolomics after sample collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Hospital of Traditional Chinese Medicine, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided